CLINICAL TRIAL: NCT03100734
Title: A Multicentre Observational Study to Evaluate the Real-Life Effectiveness of Benepali® Following Transition From Enbrel® in Patients With Rheumatoid Arthritis (RA) and Axial Spondyloarthritis (axSpA) - The BENEFIT Study
Brief Title: Observational Study to Evaluate the Real-Life Effectiveness of Benepali Following Transition From Enbrel
Acronym: BENEFIT
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Collaborators: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: EUR-BNP-16-11030
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Rheumatoid Arthritis; Axial Spondyloarthritis
Keywords: Observational; Biosimilar; Etanercept; Benepali; Enbrel
MeSH Terms: conditions — Arthritis, Rheumatoid; Axial Spondyloarthritis | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- With RA: Participants with RA previously treated with Enbrel and transitioned to Benepali
  Interventions: Biological: Benepali; Biological: Enbrel
- With axSpA: Participants with axSpA previously treated with Enbrel and transitioned to Benepali
  Interventions: Biological: Benepali; Biological: Enbrel

INTERVENTIONS:
Biological: Benepali — As specified in the treatment arm
Biological: Enbrel — As specified in the treatment arm
  Other Names: etanercept

SUMMARY:
The primary objective is to evaluate the effectiveness of Benepali in participants with Rheumatoid Arthritis (RA) and axial spondyloarthritis (axSpA), including participants with Ankylosing Spondylitis (AS) and non-radiographic axSpA, following their transition from treatment with Enbrel.

The secondary objectives of this study are to describe clinical characteristics of patients transitioned from Enbrel® to Benepali® in routine practice, to evaluate safety during and following the transition from Enbrel to Benepali and to evaluate patient-reported outcomes during and following the transition from Enbrel to Benepali.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have been diagnosed with either rheumatoid arthritis or axial spondyloarthritis, according to local practice
* Transition from Enbrel to Benepali at the physician's (Investigator's) discretion prior to enrolment into the study
* Must have been treated with the same dose of Enbrel for at least 6 months prior to transition to Benepali and have at least 1 efficacy data value including but not restricted to DAS-28 or BASDAI during that period
* Must have a stable disease throughout the 2 month prior to enrolment based on the Investigator's judgement
* Women of childbearing potential should be advised to use appropriate contraception to avoid becoming pregnant during Benepali therapy and for three weeks after discontinuation of therapy

Key Exclusion Criteria:

* Have any medical conditions that precludes administration of Benepali according to Summary of Product Characteristics (SmPC), such as the following:
* Hypersensitivity to the Benepali active substance, or to any of the associated excipients
* Sepsis, or risk of sepsis
* Active clinically significant local or chronic viral, bacterial or fungal infection, or any major episode of infection requiring hospitalization or treatment with parenteral anti-infectives within 2 months prior to enrollment
* Show any clinical sign or medical condition not allowing for treatment continuation (of etanercept) in the judgment of the Investigator
* Treatment with another biologic agent
* Are currently receiving or have previously received any therapies that would preclude administration of Benepali, such as the following:
* Immunizations with live or live-attenuated vaccines within the last 6 months prior to transition point and throughout the observation period
* Treatment with investigational agents within the last 6 months prior to transition point and during the period of observation.
* Any other unspecified reasons that would, in the opinion of the Investigator, make the patient unsuitable for enrollment.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants With Rheumatoid Arthritis or Axial Spondyloarthritis to be identified from Primary Care Practice / Hospital
Sampling Method: Probability Sample
Enrollment: 585 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Change from transition point in Disease Activity Score (DAS-28 score) | Approximately 3 months after the transition
  Score of 28 joints examined
Change from transition point in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score | Approximately 3 months after the transition
  Mean BASDAI score

SECONDARY OUTCOMES:
Change in the DAS-28 score over time from the value obtained at the Transition Point | Approximately 3 and 6 months after the transition
  Score of 28 joints examined
Proportion of participants with low disease activity or remission over time following Transition Point | Approximately 3 and 6 months after the transition
  Defined as DAS-28 score ≤ 3.2 or ≤ 2.6
Proportion of participants with worsening disease over time following Transition Point | Approximately 3 and 6 months after the transition
  Defined by an increase in DAS-28 of ≥ 1.2, and a minimum DAS score of 3.2
Proportion of participants with an improvement of ≥ 1.2 points in DAS-28 score from Transition Point | Approximately 3 and 6 months after the transition
  Improvement of ≥ 1.2 points in DAS-28 score data collected
Change in the General Health Score (assessed using VAS) over time following transition point | Approximately 3 and 6 months after the transition
  Assessed using Visual Analogue Scale (VAS) over time
Change in the BASDAI score over time from the value obtained at the Transition Point | Approximately 3 and 6 months after the transition
  BASDAI score
Change in Ankylosing Spondylitis Disease Activity Score-Erythrocyte Sedimentation Rate (ASDAS-ESR ) or C-Reactive Protein (CRP) score over time from the value obtained at the Transition Point | Approximately 3 and 6 months after the transition
  (ASDAS-ESR ) or (CRP) score
Proportion of participants with worsening disease over time following Transition Point | Approximately 3 and 6 months after the transition
  Defined by an increase in ASDAS score of ≥1.1, and a minimum ASDAS score of 2.1
Number of Participants Experiencing Adverse Events (AEs) and Serious Adverse Events (SAEs) by Severity | Approximately 3 and 6 months after the transition
  Safety surveillance
Change in Patient Global Assessment (PtGA)-Disease activity-VAS score over time from the value obtained at the Transition Point | Approximately 3 and 6 months after the transition
  Assessed using Disease activity-VAS score
Change in Patient Global Assessment - Visual Analogue Scale (PGA PAIN-VAS) score over time from the value obtained at the Transition Point | Approximately 3 and 6 months after the transition
  Assessed using PAIN-VAS score
Change in Patient PGA FATIGUE -VAS score over time from the value obtained at the Transition Point | Approximately 3 and 6 months after the transition
  Assessed using FATIGUE - VAS score
Change in Health Assessment Questionnaire Disability Index (HAQ-DI) score over time from the value obtained at the Transition Point | Approximately 3 and 6 months after the transition
  Assessed using the HAQ-DI score
Change in PAIN-VAS score over time from the value obtained at the Transition Point | Approximately 3 and 6 months after the transition
  Assessed using Pain - VAS score
Change in FATIGUE -VAS score over time from the value obtained at the Transition Point | Approximately 3 and 6 months after the transition
  Assessed using FATIGUE - VAS score
Change in HAQ-DI score over time from the value obtained at the Transition Point | Approximately 3 and 6 months after the transition
  Assessed using the HAQ-DI score
Number of Participants by Demographic Category | At baseline and approximately 3 and 6 months after the transition
Number of Participants by Relevant Medical History | At baseline and approximately 3 and 6 months after the transition
Number of Participants by Disease Status | At baseline and approximately 3 and 6 months after the transition
Number of Participants by Relevant Medication Use | At baseline and approximately 3 and 6 months after the transition

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, München, Bavaria, Germany

REFERENCES:
- See also: Manuscript description — https://www.clinexprheumatol.org/abstract.asp?a=14829